CLINICAL TRIAL: NCT04627389
Title: Esthetic Outcomes Evaluation of Unilateral Cleft Lip Repaired by Orbicularis Oris Z-plasty Modification of Modified Millard Technique Versus Modified Millard Technique. A Randomized Clinical Trail.
Brief Title: Orbicularis Oris Z-plasty Modification of Modified Millard Technique and the Esthetic Outcome of Cleft Lip Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, lecturer,oral surgery, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27/9/20
Record Dates: First submitted 2020-11-04; First posted 2020-11-13 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Cleft Lip
Keywords: cleft lip; chelioplasty; modified millard; orbicularis oris modification
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study arm (Experimental): 20 patients with a unilateral cleft lip will be repaired with orbicularis oris muscle Z-plasty modification of modified Millard technique
  Interventions: Procedure: orbicularis oris muscle Z- plasty modification of modified millard technique
- controlled arm (Active Comparator): 20 patients with a unilateral cleft lip will be repaired with modified Millard technique
  Interventions: Procedure: modified millard technique

INTERVENTIONS:
Procedure: orbicularis oris muscle Z- plasty modification of modified millard technique — After orbicularis oris muscle had been released from the overlying skin, the previously marked points using methylene blue for designing the z-plasty were shown to be followed by back-cut incisions including the OOM and inner mucosa in both medial and lateral elements without involving the overlying skin. This procedure resulted in two triangular flaps in both segments
  Arms: study arm
Procedure: modified millard technique — no z-plasty modification
  Arms: controlled arm

SUMMARY:
This study aimed to evaluate the effect of orbicularis oris muscle z-plasty modification of modified Millard technique on the esthetic outcome and length of the repaired lip

DETAILED DESCRIPTION:
forty patients with a unilateral cleft lip will be enrolled in this randomized comparative study. The patients will be divided into two groups, the control (group A) who treated with the modified Millard technique and the study group who repaired by orbicularis oris muscle Zplasty modification of modified Millard technique (group B).

ELIGIBILITY:
Inclusion Criteria:

* non-syndromic cleft lip patients.
* Primary, unilateral, complete or incomplete cleft lip.
* The patient's age is younger than six months.
* lip repair performed by one craniofacial surgeon

Exclusion Criteria

* syndromic cleft lip.
* Secondary lip treatment (previously operated cases)
* Bilateral cleft lip
* Patients are older than six months. Associated Cardiac anomalies. Any systemic condition

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
lip legth | immediate postoperative
  evaluate the lip length of the cleft side changes from preoperative at immediate postoperative

SECONDARY OUTCOMES:
Philtral ridge length symmetry index assessment | 6months
  Philtral ridge symmetry index was calculated as follow:- (philtral ridge length by mm at cleft side)/(philtral ridge length by mm at non-clefted side)×100
Scar width assessment by photograph | 6months
  Standard photography was taken; objective measurements were obtained from the photographs using the ruler as a control reference.
  One standard surgical ruler was placed over the lower lip and a frontally orientated photograph of the patient was taken at 6m follow up to assess scar width using the Image J1.5i0R program. The first point was 1mm above the white roll and the second point was 1mm below the C-flap suture line . Scar width will be measured by two assessors and the mean score of two assessors was calculated
scar width by ultrasound | 6months
  scar width will be quantified by ultrasound. The transducer placement with its upper border touching the columella-philtral junction, upper lip imaging obtained and the scar width will be measured.
scar elascitity | 6months
  Scar elasticity will be quantified by ultrasound. The transducer, coupled with several millimeters of ultrasound gel, was smoothly placed in the longitudinal section and perpendicular to the skin without compressing the tissue. Compare scar stiffness in relation to adjacent normal tissue

CONTACTS AND LOCATIONS:
Overall Officials: shaimaa refahee, phd, Principal Investigator — Fayoum University
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No